CLINICAL TRIAL: NCT05022472
Title: Project 2VIDA! SARS-CoV-2 Vaccine Intervention Delivery for Adults in Southern California
Brief Title: Project 2VIDA! COVID-19 Vaccine Intervention Delivery for Adults in Southern California
Acronym: 2VIDA!
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Britt Skaathun (Other)
Collaborators: San Ysidro Health Center (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor-Investigator, Britt Skaathun, Assistant Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 210630S; 1R01MD016872-01 (NIH)
Record Dates: First submitted 2021-08-18; First posted 2021-08-26 (Actual); Results first posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Vaccine Refusal; Covid19
Keywords: Latinx; African American; COVID-19; Community-based participatory research
MeSH Terms: conditions — Vaccination Refusal; COVID-19 | interventions — Educational Status; Health Promotion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention (Experimental): We will use a 2-armed randomized controlled trial (RCT) where Latino and AA adults >18 years or older from six participating communities and surrounding community health centers (CHC) will be assigned to the 2 VIDA! intervention (n=3 CHC; N=500 participants) or to the control site (e.g., standard of care) (n=3 CHC; N=500 participants). The two major components of the 2VIDA! intervention are: COVID-19 Individual Awareness and Education, COVID-19 Community Outreach and Health Promotion, COVID-19 Individual Health Education and Linkages to Medical and Supportive Services, and pop-up vaccination stations in Latino and AA communities.
  Interventions: Behavioral: COVID-19 Individual Awareness and Education.; Behavioral: COVID-19 Community Outreach & Health Promotion.; Behavioral: COVID-19 Individual Health Education & Linkages to Medical and Supportive Services.; Biological: Pop-up community vaccination sites
- Standard of care (No Intervention): The standard of care for vaccine delivery at the control sites. This includes individuals who make an appointment on their own or receive the vaccine at a health center and may receive information about the vaccine from their primary healthcare provider.

INTERVENTIONS:
Behavioral: COVID-19 Individual Awareness and Education. — The 2VIDA! working group has developed culturally competent COVID-19 educational and outreach materials (available printed and electronically) in English and Spanish that are written at the 8th grade level (the average reading level of adults in the United States) that peer-health educators will distributed to community members during their visits to the participating SYH community centers, door-to-door, local supermarkets, and CBO's in the selected communities. These materials have general information on COVID-19 as well as educational information and resources regarding COVID-19 prevention, symptoms, testing, contact tracing, COVID-19 vaccine (how it works, technology used, administration [2-dose series and importance of vaccine completion]), safety concerns, benefits, dispelling common misconceptions and misinformation, and other topics identified based on community needs. This information will be updated monthly to ensure the most up to date information.
  Arms: Intervention
Behavioral: COVID-19 Community Outreach & Health Promotion. — Peer-health educators will work with local CBO's and facilitate a combination of live broadcast sessions, pre-recorded webinars, social media posts, and other outreach activities in English and Spanish reaching community members with information on the above COVID-19 related topics as well as other identified needs such as what to do if a family member is infected and where you can get the COVID-19 vaccine. The goal is to reach 10,000 viewers (per session) in the various social media platforms in the three randomly selected communities.
  Arms: Intervention
Behavioral: COVID-19 Individual Health Education & Linkages to Medical and Supportive Services. — SYHealth will establish a COVID-19 Resource Center within the participating health centers in the three randomly selected communities (intervention sites only) providing individual COVID-19 related health education and linkages to medical and supportive services for patients and community members in need of additional education and support regarding COVID-19 disease and COVID-19 vaccine.
  Arms: Intervention
Biological: Pop-up community vaccination sites — We will offer the COVID-19 vaccine at the participating SYHealth community health centers and pop-up vaccination stations that will be set-up in these communities (intervention sites) as part of the interventions efforts to increase access and uptake of the COVID-19 vaccine. We have identified various open spaces (e.g., public parks) in these communities to set-up the vaccination stations. Additionally, data will be collected to assess individual, social, and contextual factors related to access, acceptance, and uptake of the COVID-19 vaccine.The survey will last approximately 10-15 minutes and will be self-administered in both English and Spanish. Following the survey participants will be offered the COVID-19 vaccine and will be made an automatic appointment for the 2nd dose (4-week follow-up) and will be asked to complete a 5 min survey during the follow-up visit.
  Arms: Intervention

SUMMARY:
The United States (U.S.) is the country with the largest number of infections and deaths due to COVID- 19 and racial/ethnic minorities are disproportionately affected. Acceptance and uptake of COVID-19 vaccines will be instrumental to ending the pandemic. To this end, 2VIDA! (SARS-CoV-2 Vaccine Intervention Delivery for Adults in Southern California) is a multilevel intervention to address individual, social, and contextual factors related to access to, and acceptance of, the COVID-19 vaccine by implementing and assessing a COVID-19 vaccination protocol among Latino and African American (AA) adults (>18 years old) in San Diego. 2VIDA! builds on our previous CBPR efforts and centers on conducting COVID-19 Individual awareness and education, linkages to medical and supportive services, and Community Outreach and Health Promotion in the intervention sites (Phase 1); and offering the COVID-19 vaccine to Latino and AA adults (>18 years old) in federally-qualified health centers and pop-up vaccination stations in communities highly impacted by the pandemic and identifying individual and structural barriers to COVID-19 immunization (Phase 2).

DETAILED DESCRIPTION:
As of January 2021, the World Health Organization (WHO) reports that 89 million cases of COVID-19 (SARS- CoV-2) have been confirmed and have resulted in more than 1.9 million deaths globally. Currently, the United States (U.S.) is the country with the largest number of infections and deaths due to COVID-19, with a total of 22 million infections and 373,167 deaths. Furthermore, early findings that have examined COVID-19 demographics show that racial and ethnic minorities in the U.S. are bearing a disproportionate number of COVID-19 cases and deaths irrespective of geographic region. While there's no evidence that people of color (POC) have genetic or biological factors that make them more likely to be affected by COVID-19, they are more likely to have underlying health conditions, live in multi-generational homes, live in densely populated areas, have limited access to healthcare, and have jobs that are considered essential and involve interaction with the public. All of these factors contribute to higher rates of infection and adverse outcomes due to COVID-19. Although COVID-19 preventive behaviors such as hand washing, mask wearing, and social distancing have been shown to be effective in curbing the spread of the virus, acceptance and uptake of COVID-19 vaccines will be instrumental to ending the pandemic. However, public confidence in vaccination is fragile, especially among racial and ethnic minorities. To this end, we have formed an intervention working group comprised of representatives from community and academic organizations to address challenges in COVID-19 vaccination uptake among Latino and African American (AA) communities in Southern California by using a community-based participatory research (CBPR) approach. Project 2VIDA! (SARS-CoV-2 Vaccine Intervention Delivery for Adults in Southern California), is a multilevel intervention to address individual, social, and contextual factors related to access to, and acceptance of, the COVID-19 vaccine among Latino and AA adults (>18 years old) across six highly affected communities in Southeast San Diego. 2VIDA! seeks to implement and assess a COVID-19 vaccination protocol to increase interest and uptake of COVID-19 vaccine, provide COVID-19 vaccines in the community, and establish a model for the rapid vaccination of Latino and AA adults that could be generalizable to other highly affected communities. 2VIDA! builds on our previous CBPR efforts and centers on conducting COVID-19 community outreach and health promotion, Individual awareness and education, and linkages to medical and supportive services and offering the COVID-19 vaccine to Latino and AA adults (>18 years old) in community health centers (CHC) and mini-vaccination stations in communities highly impacted by the pandemic in San Diego County.

ELIGIBILITY:
Inclusion Criteria:

* age 16 years or older
* identify as Latinx and/or AA
* biologically male or female
* be a resident of one of the six communities selected for this study (National City, Lincoln Park, Logan Heights, Valencia Park, Chula Vista or San Ysidro)
* literate in English or Spanish
* no known history of severe allergic reactions to any components of the vaccine
* no history of immune disease
* not be pregnant
* no plans to move from the area in the following 30 days
* able to provide voluntary informed consent
* able to provide complete contact information for themselves and two additional contact individuals (for follow-up 2nd vaccine shot)

Exclusion Criteria:

* under 16 years old
* pregnant women
* individuals unable to consent

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1051 (Actual)
Dates: Start 2021-07-16 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Argentina E Servin, MD,MPH, Principal Investigator — UC San Diego
Locations (6):
- United States (6):
  - San Ysidro Health Chula Vista, Chula Vista, California
  - Care View Health Center, San Diego, California
  - San Ysidro Health Care View Health Center, San Diego, California
  - San Ysidro Health Euclid, San Diego, California
  - San Ysidro Health King-Chavez Health Center, San Diego, California
  - San Ysidro Health, San Ysidro, California

REFERENCES:
- [Derived] Skaathun B, Salgin L, Munoz FA, Talavera GA, Smith DM, Stockman JK, O'Bryan SE, Ramirez D, James-Price C, Servin AE. Study protocol: Project 2VIDA! SARS-CoV-2 vaccine intervention delivery for adults in Southern California. Front Public Health. 2024 Mar 14;12:1291332. doi: 10.3389/fpubh.2024.1291332. eCollection 2024. PMID 38550328

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: We conducted a 2-armed randomized controlled trial (RCT) with 1,051 Latino and African American adults (≥18 years) from six communities and affiliated community health centers (CHCs). Participants were randomized to either the 2VIDA! intervention group (n=517; 3 CHCs) or control (standard of care; n=534; 3 CHCs).
  The 2VIDA! intervention included four components: (1) COVID-19 Individual Awareness and Education, (2) COVID-19 Community Outreach and Health Promotion, (3) Individual Health Education and Linkages to Services, and (4) Pop-up Vaccination Stations.
  COVID-19 Individual Awareness & Education: Peer-health educators distributed culturally competent, bilingual (English/Spanish) COVID-19 materials at community centers, door-to-door, local markets, and CBOs. Materials covered prevention, symptoms, testing, vaccines, and debunking myths, and were updated monthly.
  Community Outreach & Health Promotion: Educators partnered with CBOs to deliver live sessions, webinars, and social media outreach on COVID-19 topics, aiming to reach 10,000 viewers per session in each intervention community.
  Individual Health Education & Linkages: COVID-19 Resource Centers were set up at intervention CHCs to offer personalized education and referrals to medical/support services.
  Pop-up Vaccination Sites: COVID-19 vaccines were offered at CHCs and temporary community sites in intervention areas to improve access and uptake.
Period: Overall Study
Arm/Group | Intervention | Standard of Care
Started | 517 | 534
Completed | 339 | 435
Not Completed | 178 | 99

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Standard of Care | Total
Number analyzed (Participants) | 517 | 534 | 1051
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 3 | 4
  Between 18 and 65 years | 449 | 382 | 831
  >=65 years | 67 | 149 | 216
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (16.9) | 52.7 (17.4) | 48.2 (17.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 2 participants refused to answer in the standard of care group.
  Participants
    Sex: number analyzed (Participants) | 517 | 532 | 1049
    Sex: Female | 272 | 358 | 630
    Sex: Male | 245 | 174 | 419
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: AI/AN/Asian/NH/PI | 6 | 11 | 17
  Race/Ethnicity: Black or African American | 34 | 29 | 63
  Race/Ethnicity: Hispanic or Latino/a | 460 | 475 | 935
  Race/Ethnicity: White | 5 | 10 | 15
  Race/Ethnicity: Multiracial | 8 | 7 | 15
  Race/Ethnicity: Don't know/Refuse to answer | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 517 | 534 | 1051

OUTCOME MEASURES:

1. Primary Outcome: Change in Vaccine Hesitancy
Description: Based on the definition of the Strategic Advisory Group of Experts (SAGE) Working Group on Vaccine Hesitancy (WG), hesitancy refers to "delay in acceptance or refusal of vaccination despite availability of vaccination services. Vaccine hesitancy is complex and context specific, varying across time, place and vaccines. It is influenced by factors such as complacency, convenience and confidence."
Time Frame: Baseline (current), and follow-up (4-weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 339 | 435
Participants
  Baseline: I believe a vaccine can help control the spread of COVID-19: Agree | 282 | 387
  Baseline: I believe a vaccine can help control the spread of COVID-19: Disagree or Neutral | 57 | 48
  Baseline: I believe a vaccine can help control the spread of COVID-19: Yes | 0 | 0
  Baseline: I believe a vaccine can help control the spread of COVID-19: No | 0 | 0
  Follow-up: I believe a vaccine can help control the spread of COVID-19: Agree | 274 | 366
  Follow-up: I believe a vaccine can help control the spread of COVID-19: Disagree or Neutral | 65 | 69
  Follow-up: I believe a vaccine can help control the spread of COVID-19: Yes | 0 | 0
  Follow-up: I believe a vaccine can help control the spread of COVID-19: No | 0 | 0
  Baseline: If I knew I had been infected with COVID-19 before, I would not get the vaccine.: Agree | 61 | 85
  Baseline: If I knew I had been infected with COVID-19 before, I would not get the vaccine.: Disagree or Neutral | 278 | 350
  Baseline: If I knew I had been infected with COVID-19 before, I would not get the vaccine.: Yes | 0 | 0
  Baseline: If I knew I had been infected with COVID-19 before, I would not get the vaccine.: No | 0 | 0
  Follow-up: If I knew I had been infected with COVID-19 before, I would not get the vaccine.: Agree | 50 | 54
  Follow-up: If I knew I had been infected with COVID-19 before, I would not get the vaccine.: Disagree or Neutral | 289 | 381
  Follow-up: If I knew I had been infected with COVID-19 before, I would not get the vaccine.: Yes | 0 | 0
  Follow-up: If I knew I had been infected with COVID-19 before, I would not get the vaccine.: No | 0 | 0
  Baseline: When everyone else is vaccinated against COVID-19, then I don't have to get vaccinated.: Agree | 34 | 46
  Baseline: When everyone else is vaccinated against COVID-19, then I don't have to get vaccinated.: Disagree or Neutral | 305 | 389
  Baseline: When everyone else is vaccinated against COVID-19, then I don't have to get vaccinated.: Yes | 0 | 0
  Baseline: When everyone else is vaccinated against COVID-19, then I don't have to get vaccinated.: No | 0 | 0
  Follow-up: When everyone else is vaccinated against COVID-19, then I don't have to get vaccinated.: Agree | 34 | 32
  Follow-up: When everyone else is vaccinated against COVID-19, then I don't have to get vaccinated.: Disagree or Neutral | 305 | 403
  Follow-up: When everyone else is vaccinated against COVID-19, then I don't have to get vaccinated.: Yes | 0 | 0
  Follow-up: When everyone else is vaccinated against COVID-19, then I don't have to get vaccinated.: No | 0 | 0
  (Baseline) The country where the COVID-19 vaccine is made affects my decision to get vaccinated.: Agree | 0 | 0
  (Baseline) The country where the COVID-19 vaccine is made affects my decision to get vaccinated.: Disagree or Neutral | 0 | 0
  (Baseline) The country where the COVID-19 vaccine is made affects my decision to get vaccinated.: Yes | 65 | 51
  (Baseline) The country where the COVID-19 vaccine is made affects my decision to get vaccinated.: No | 274 | 384
  (Follow-up) The country where the COVID-19 vaccine is made affects my decision to get vaccinated.: Agree | 0 | 0
  (Follow-up) The country where the COVID-19 vaccine is made affects my decision to get vaccinated.: Disagree or Neutral | 0 | 0
  (Follow-up) The country where the COVID-19 vaccine is made affects my decision to get vaccinated.: Yes | 57 | 54
  (Follow-up) The country where the COVID-19 vaccine is made affects my decision to get vaccinated.: No | 282 | 381
  (Baseline) My decision to get the COVID-19 vaccine depends on my family doctor's recommendation: Agree | 0 | 0
  (Baseline) My decision to get the COVID-19 vaccine depends on my family doctor's recommendation: Disagree or Neutral | 0 | 0
  (Baseline) My decision to get the COVID-19 vaccine depends on my family doctor's recommendation: Yes | 131 | 220
  (Baseline) My decision to get the COVID-19 vaccine depends on my family doctor's recommendation: No | 208 | 215
  (Follow-up) My decision to get the COVID-19 vaccine depends on my family doctor's recommendation: Agree | 0 | 0
  (Follow-up) My decision to get the COVID-19 vaccine depends on my family doctor's recommendation: Disagree or Neutral | 0 | 0
  (Follow-up) My decision to get the COVID-19 vaccine depends on my family doctor's recommendation: Yes | 153 | 259
  (Follow-up) My decision to get the COVID-19 vaccine depends on my family doctor's recommendation: No | 186 | 176
  (Baseline) My decision to get the COVID-19 vaccine depends on Health Department guidance: Agree | 0 | 0
  (Baseline) My decision to get the COVID-19 vaccine depends on Health Department guidance: Disagree or Neutral | 0 | 0
  (Baseline) My decision to get the COVID-19 vaccine depends on Health Department guidance: Yes | 165 | 157
  (Baseline) My decision to get the COVID-19 vaccine depends on Health Department guidance: No | 174 | 278
  (Follow-up) My decision to get the COVID-19 vaccine depends on Health Department guidance: Agree | 0 | 0
  (Follow-up) My decision to get the COVID-19 vaccine depends on Health Department guidance: Disagree or Neutral | 0 | 0
  (Follow-up) My decision to get the COVID-19 vaccine depends on Health Department guidance: Yes | 186 | 204
  (Follow-up) My decision to get the COVID-19 vaccine depends on Health Department guidance: No | 153 | 231
  (Baseline) My decision to get the COVID-19 vaccine depends on proven long-term safety: Agree | 0 | 0
  (Baseline) My decision to get the COVID-19 vaccine depends on proven long-term safety: Disagree or Neutral | 0 | 0
  (Baseline) My decision to get the COVID-19 vaccine depends on proven long-term safety: Yes | 83 | 72
  (Baseline) My decision to get the COVID-19 vaccine depends on proven long-term safety: No | 256 | 363
  (Follow-up) My decision to get the COVID-19 vaccine depends on proven long-term safety: Agree | 0 | 0
  (Follow-up) My decision to get the COVID-19 vaccine depends on proven long-term safety: Disagree or Neutral | 0 | 0
  (Follow-up) My decision to get the COVID-19 vaccine depends on proven long-term safety: Yes | 86 | 85
  (Follow-up) My decision to get the COVID-19 vaccine depends on proven long-term safety: No | 253 | 350
  (Baseline) My decision to get the COVID-19 vaccine depends on its use in other countries.: Agree | 0 | 0
  (Baseline) My decision to get the COVID-19 vaccine depends on its use in other countries.: Disagree or Neutral | 0 | 0
  (Baseline) My decision to get the COVID-19 vaccine depends on its use in other countries.: Yes | 38 | 28
  (Baseline) My decision to get the COVID-19 vaccine depends on its use in other countries.: No | 301 | 407
  (Follow-up) My decision to get the COVID-19 vaccine depends on its use in other countries.: Agree | 0 | 0
  (Follow-up) My decision to get the COVID-19 vaccine depends on its use in other countries.: Disagree or Neutral | 0 | 0
  (Follow-up) My decision to get the COVID-19 vaccine depends on its use in other countries.: Yes | 36 | 52
  (Follow-up) My decision to get the COVID-19 vaccine depends on its use in other countries.: No | 303 | 383
  (Baseline) My decision to get the COVID-19 vaccine depends on my risk of infection at the time: Agree | 0 | 0
  (Baseline) My decision to get the COVID-19 vaccine depends on my risk of infection at the time: Disagree or Neutral | 0 | 0
  (Baseline) My decision to get the COVID-19 vaccine depends on my risk of infection at the time: Yes | 83 | 119
  (Baseline) My decision to get the COVID-19 vaccine depends on my risk of infection at the time: No | 256 | 316
  (Follow-up) My decision to get the COVID-19 vaccine depends on my risk of infection at the time: Agree | 0 | 0
  (Follow-up) My decision to get the COVID-19 vaccine depends on my risk of infection at the time: Disagree or Neutral | 0 | 0
  (Follow-up) My decision to get the COVID-19 vaccine depends on my risk of infection at the time: Yes | 75 | 117
  (Follow-up) My decision to get the COVID-19 vaccine depends on my risk of infection at the time: No | 264 | 318
  (Baseline) My decision to get the COVID-19 vaccine depends on how easy it is to access.: Agree | 0 | 0
  (Baseline) My decision to get the COVID-19 vaccine depends on how easy it is to access.: Disagree or Neutral | 0 | 0
  (Baseline) My decision to get the COVID-19 vaccine depends on how easy it is to access.: Yes | 100 | 80
  (Baseline) My decision to get the COVID-19 vaccine depends on how easy it is to access.: No | 239 | 355
  (Follow-up) My decision to get the COVID-19 vaccine depends on how easy it is to access.: Agree | 0 | 0
  (Follow-up) My decision to get the COVID-19 vaccine depends on how easy it is to access.: Disagree or Neutral | 0 | 0
  (Follow-up) My decision to get the COVID-19 vaccine depends on how easy it is to access.: Yes | 104 | 109
  (Follow-up) My decision to get the COVID-19 vaccine depends on how easy it is to access.: No | 235 | 326
  (Baseline) My decision to get the COVID-19 vaccine depends on whether it's free of charge: Agree | 0 | 0
  (Baseline) My decision to get the COVID-19 vaccine depends on whether it's free of charge: Disagree or Neutral | 0 | 0
  (Baseline) My decision to get the COVID-19 vaccine depends on whether it's free of charge: Yes | 109 | 112
  (Baseline) My decision to get the COVID-19 vaccine depends on whether it's free of charge: No | 230 | 323
  (Follow-up) My decision to get the COVID-19 vaccine depends on whether it's free of charge: Agree | 0 | 0
  (Follow-up) My decision to get the COVID-19 vaccine depends on whether it's free of charge: Disagree or Neutral | 0 | 0
  (Follow-up) My decision to get the COVID-19 vaccine depends on whether it's free of charge: Yes | 125 | 126
  (Follow-up) My decision to get the COVID-19 vaccine depends on whether it's free of charge: No | 214 | 309
  (Baseline) My decision depends on whether vaccines help end movement and gathering limits: Agree | 0 | 0
  (Baseline) My decision depends on whether vaccines help end movement and gathering limits: Disagree or Neutral | 0 | 0
  (Baseline) My decision depends on whether vaccines help end movement and gathering limits: Yes | 41 | 37
  (Baseline) My decision depends on whether vaccines help end movement and gathering limits: No | 298 | 398
  (Follow-up) My decision depends on whether vaccines help end movement and gathering limits: Agree | 0 | 0
  (Follow-up) My decision depends on whether vaccines help end movement and gathering limits: Disagree or Neutral | 0 | 0
  (Follow-up) My decision depends on whether vaccines help end movement and gathering limits: Yes | 58 | 65
  (Follow-up) My decision depends on whether vaccines help end movement and gathering limits: No | 281 | 370
  (Baseline) My decision to get the COVID-19 vaccine depends on other factors (please specify): Agree | 0 | 0
  (Baseline) My decision to get the COVID-19 vaccine depends on other factors (please specify): Disagree or Neutral | 0 | 0
  (Baseline) My decision to get the COVID-19 vaccine depends on other factors (please specify): Yes | 28 | 27
  (Baseline) My decision to get the COVID-19 vaccine depends on other factors (please specify): No | 311 | 408
  (Follow-up) My decision to get the COVID-19 vaccine depends on other factors (please specify): Agree | 0 | 0
  (Follow-up) My decision to get the COVID-19 vaccine depends on other factors (please specify): Disagree or Neutral | 0 | 0
  (Follow-up) My decision to get the COVID-19 vaccine depends on other factors (please specify): Yes | 36 | 51
  (Follow-up) My decision to get the COVID-19 vaccine depends on other factors (please specify): No | 303 | 384

2. Secondary Outcome: Change in Health Literacy
Description: Assessment of ease/difficulty in finding information on symptoms, finding out what to do if infected, understand what authorities say, judge reliability of information, follow recommendations, decide on prevention behaviors. (Adapted from the WHO COVID-19 Survey Tool and Guidance).
Time Frame: Baseline and follow-up (4-weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 339 | 435
Participants
  (Baseline) How easy is it to find the COVID-19 information you need?: Easy | 258 | 323
  (Baseline) How easy is it to find the COVID-19 information you need?: Difficult or Neutral | 81 | 112
  (Follow-up) How easy is it to find the COVID-19 information you need?: Easy | 265 | 337
  (Follow-up) How easy is it to find the COVID-19 information you need?: Difficult or Neutral | 74 | 98
  (Baseline) How easy is it to understand what to do if you think you have COVID-19?: Easy | 244 | 309
  (Baseline) How easy is it to understand what to do if you think you have COVID-19?: Difficult or Neutral | 95 | 126
  (Follow-up) How easy is it to understand what to do if you think you have COVID-19?: Easy | 254 | 337
  (Follow-up) How easy is it to understand what to do if you think you have COVID-19?: Difficult or Neutral | 85 | 98
  (Baseline) How easy is it to judge if COVID-19 info in the media is reliable?: Easy | 146 | 224
  (Baseline) How easy is it to judge if COVID-19 info in the media is reliable?: Difficult or Neutral | 193 | 211
  (Follow-up) How easy is it to judge if COVID-19 info in the media is reliable?: Easy | 174 | 223
  (Follow-up) How easy is it to judge if COVID-19 info in the media is reliable?: Difficult or Neutral | 165 | 212
  (Baseline) How easy is it to understand COVID-19 rules and recommendations from authorities?: Easy | 241 | 318
  (Baseline) How easy is it to understand COVID-19 rules and recommendations from authorities?: Difficult or Neutral | 98 | 117
  (Follow-up) How easy is it to understand COVID-19 rules and recommendations from authorities?: Easy | 266 | 350
  (Follow-up) How easy is it to understand COVID-19 rules and recommendations from authorities?: Difficult or Neutral | 73 | 85
  (Baseline) How easy is it to follow recommendations to protect yourself from COVID-19?: Easy | 278 | 355
  (Baseline) How easy is it to follow recommendations to protect yourself from COVID-19?: Difficult or Neutral | 61 | 80
  (Follow-up) How easy is it to follow recommendations to protect yourself from COVID-19?: Easy | 274 | 372
  (Follow-up) How easy is it to follow recommendations to protect yourself from COVID-19?: Difficult or Neutral | 65 | 63
  (Baseline) How easy is it to understand when to stay home from work or school due to COVID-19?: Easy | 266 | 357
  (Baseline) How easy is it to understand when to stay home from work or school due to COVID-19?: Difficult or Neutral | 73 | 78
  (Follow-up) How easy is it to understand when to stay home from work or school due to COVID-19?: Easy | 277 | 365
  (Follow-up) How easy is it to understand when to stay home from work or school due to COVID-19?: Difficult or Neutral | 62 | 70
  (Baseline) How easy is it to follow recommendations on when to stay home from work or school?: Easy | 251 | 341
  (Baseline) How easy is it to follow recommendations on when to stay home from work or school?: Difficult or Neutral | 88 | 94
  (Follow-up) How easy is it to follow recommendations on when to stay home from work or school?: Easy | 265 | 356
  (Follow-up) How easy is it to follow recommendations on when to stay home from work or school?: Difficult or Neutral | 74 | 79
  (Baseline) How easy is it to understand when to engage in social activities or avoid them?: Easy | 271 | 351
  (Baseline) How easy is it to understand when to engage in social activities or avoid them?: Difficult or Neutral | 68 | 84
  (Follow-up) How easy is it to understand when to engage in social activities or avoid them?: Easy | 280 | 360
  (Follow-up) How easy is it to understand when to engage in social activities or avoid them?: Difficult or Neutral | 59 | 75
  (Baseline) How easy is it to follow advice on when to engage in or avoid social activities?: Easy | 261 | 341
  (Baseline) How easy is it to follow advice on when to engage in or avoid social activities?: Difficult or Neutral | 78 | 94
  (Follow-up) How easy is it to follow advice on when to engage in or avoid social activities?: Easy | 269 | 355
  (Follow-up) How easy is it to follow advice on when to engage in or avoid social activities?: Difficult or Neutral | 70 | 80

3. Secondary Outcome: Change in COVID-19 Risk Perception (Probability and Severity)
Description: Self-assessed probability and susceptibility to of contracting COVID-19 and self-assessed severity in case of contracting COVID-19. (Adapted from the WHO COVID-19 Survey Tool and Guidance).
Time Frame: Baseline and follow-up (4-weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 339 | 435
Participants
  (Baseline) How likely do you think are your chances of getting sick with COVID-19?: Likely | 160 | 222
  (Baseline) How likely do you think are your chances of getting sick with COVID-19?: Unlikely or Neutral | 179 | 213
  (Baseline) How likely do you think are your chances of getting sick with COVID-19?: Severe | 0 | 0
  (Baseline) How likely do you think are your chances of getting sick with COVID-19?: Not severe or Neutral | 0 | 0
  (Follow-up) How likely do you think are your chances of getting sick with COVID-19?: Likely | 165 | 200
  (Follow-up) How likely do you think are your chances of getting sick with COVID-19?: Unlikely or Neutral | 174 | 235
  (Follow-up) How likely do you think are your chances of getting sick with COVID-19?: Severe | 0 | 0
  (Follow-up) How likely do you think are your chances of getting sick with COVID-19?: Not severe or Neutral | 0 | 0
  (Baseline) How seriously sick do you think you will be if you got COVID-19?: Likely | 0 | 0
  (Baseline) How seriously sick do you think you will be if you got COVID-19?: Unlikely or Neutral | 0 | 0
  (Baseline) How seriously sick do you think you will be if you got COVID-19?: Severe | 54 | 87
  (Baseline) How seriously sick do you think you will be if you got COVID-19?: Not severe or Neutral | 285 | 348
  (Follow-up) How seriously sick do you think you will be if you got COVID-19?: Likely | 0 | 0
  (Follow-up) How seriously sick do you think you will be if you got COVID-19?: Unlikely or Neutral | 0 | 0
  (Follow-up) How seriously sick do you think you will be if you got COVID-19?: Severe | 57 | 87
  (Follow-up) How seriously sick do you think you will be if you got COVID-19?: Not severe or Neutral | 282 | 348

4. Secondary Outcome: Change in Preparedness and Perceived Self-efficacy
Description: Self-assessed COVID-19 self-protection and avoidance ability. (Adapted from the WHO COVID-19 Survey Tool and Guidance).
Time Frame: Baseline and follow-up (4-weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 339 | 435
Participants
  (Baseline) I feel that avoiding an infection with COVID-19 in the current situation is…: Easy | 161 | 238
  (Baseline) I feel that avoiding an infection with COVID-19 in the current situation is…: Difficult or Neutral | 178 | 197
  (Baseline) I feel that avoiding an infection with COVID-19 in the current situation is…: Very much | 0 | 0
  (Baseline) I feel that avoiding an infection with COVID-19 in the current situation is…: Not very much or at all | 0 | 0
  (Follow-up) I feel that avoiding an infection with COVID-19 in the current situation is…: Easy | 161 | 257
  (Follow-up) I feel that avoiding an infection with COVID-19 in the current situation is…: Difficult or Neutral | 178 | 178
  (Follow-up) I feel that avoiding an infection with COVID-19 in the current situation is…: Very much | 0 | 0
  (Follow-up) I feel that avoiding an infection with COVID-19 in the current situation is…: Not very much or at all | 0 | 0
  (Baseline) I know how to protect myself from coronavirus: Easy | 0 | 0
  (Baseline) I know how to protect myself from coronavirus: Difficult or Neutral | 0 | 0
  (Baseline) I know how to protect myself from coronavirus: Very much | 249 | 306
  (Baseline) I know how to protect myself from coronavirus: Not very much or at all | 90 | 129
  (Follow-up) I know how to protect myself from coronavirus: Easy | 0 | 0
  (Follow-up) I know how to protect myself from coronavirus: Difficult or Neutral | 0 | 0
  (Follow-up) I know how to protect myself from coronavirus: Very much | 245 | 320
  (Follow-up) I know how to protect myself from coronavirus: Not very much or at all | 94 | 115

5. Secondary Outcome: Access to Health Care and Utilization
Description: Type of insurance was assessed. (Adapted from the National Health Interview Survey 2020)
Time Frame: Baseline (current)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 339 | 435
Participants
  Government Funding | 126 | 339
  Private insurance (through your work)/Parents | 80 | 42
  Self-pay, out of pocket/I don't have any type of health insurance | 120 | 47
  Other/Don't know/Refuse to answer | 13 | 7

6. Secondary Outcome: Health History
Description: History of having medical conditions that could exacerbate COVID-19 infection including: type 1 and type 2 diabetes mellitus, hypertension, heart conditions (e.g., coronary artery disease), obesity (e.g., body mass index of 30kg/m2 or higher but <40km/m2), severe obesity (e.g., BMI >40 kg/m2), asthma, chronic obstructive pulmonary disease (COPD), smoking.
  "Ever told by a medical provider they had a chronic illness"
Time Frame: Baseline
Population: Ever told by a medical provider they had a chronic illness
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 339 | 435
Participants
  Yes | 161 | 320
  No | 149 | 97
  Don't know/Refuse to answer | 29 | 18

7. Other Pre Specified Outcome: Affect
Description: Affect related to COVID-19 including: close, spreading, constant, fear-inducing, media hyped, helpless, stressful, etc. (Adapted from the WHO COVID-19 Survey Tool and Guidance).
  From "Close to me" (0) to "Far away from me" (7) From "Spreading slowly" (0) to "Spreading fast" (7) From "Something I think about all the time" (0) to "Something I almost never think about" (7) From "Fear-inducing" (0) to "Not fear-inducing" (7) From "Media hyped" (0) "Not media hyped" (7) From "Something that makes me feel helpless" (0) to "Something I am able to combat with my own action" (7) From "Stressful" (0) to "Not stressful" (7)
  "Please drag and drop the slider to the statements below that best represents how you feel. There are no right or wrong answers. COVID-19 to me feels:"
Time Frame: Baseline and follow-up (4-weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 339 | 435
units on a scale
  Baseline: Close to me (0-7) Far away from me | 3.9 (2.1) | 4.2 (2.3)
  Baseline: Spreading slowly (0-7) Spreading fast | 4.5 (2.0) | 4.6 (2.1)
  Baseline: Always on my mind (0-7) Rarely on my mind | 3.9 (2.1) | 4.3 (2.1)
  Baseline: Fear-inducing (0-7) Not fear-inducing | 3.7 (2.2) | 4.1 (2.2)
  Baseline: Media hyped (0-7) Not media hyped | 4.0 (2.1) | 4.2 (2.1)
  Baseline: Makes me feel helpless (0-7) I can combat it with my actions | 4.5 (2.0) | 4.7 (2.0)
  Baseline: Stressful (0-7) Not stressful | 3.4 (2.3) | 4.1 (2.3)
  Follow-up: Close to me (0-7) Far away from me | 4.2 (2.0) | 4.6 (1.9)
  Follow-up: Spreading slowly (0-7) Spreading fast | 4.4 (1.9) | 4.5 (2.0)
  Follow-up: Something I think about all the time (0-7) Something I almost never think about | 4.3 (1.8) | 4.7 (1.9)
  Follow-up: Fear-inducing (0-7) Not fear-inducing | 4.1 (2.0) | 4.4 (2.0)
  Follow-up: Media hyped (0-7) Not media hyped | 4.3 (1.9) | 4.3 (1.9)
  Follow-up: Feel helpless (0-7) Can act to combat it | 4.8 (1.8) | 4.9 (1.7)
  Follow-up: Stressful (0-7) Not stressful | 4.0 (2.1) | 4.3 (2.2)

8. Other Pre Specified Outcome: Use of Sources of Information
Description: Use of information sources including television, newspaper, health workers, social media, radio, health department, Centers for Disease Control and Prevention (CDC), hotlines, official websites, and celebrities. (Adapted from the WHO COVID-19 Survey Tool and Guidance).
  "How often do you use the following sources for information about COVID-19?"
Time Frame: Baseline and follow-up (4-weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 339 | 435
Participants
  Baseline: Television: Often | 127 | 211
  Baseline: Television: Not often or never | 212 | 224
  Baseline: Newspapers: Often | 49 | 60
  Baseline: Newspapers: Not often or never | 290 | 375
  Baseline: Health Workers: Often | 189 | 291
  Baseline: Health Workers: Not often or never | 150 | 144
  Baseline: Socia Media: Often | 96 | 114
  Baseline: Socia Media: Not often or never | 243 | 321
  Baseline: Radio: Often | 89 | 87
  Baseline: Radio: Not often or never | 250 | 348
  Baseline: Health department: Often | 204 | 270
  Baseline: Health department: Not often or never | 135 | 165
  Baseline: CDC: Often | 190 | 250
  Baseline: CDC: Not often or never | 149 | 185
  Baseline: Celebrities or social media influencers: Often | 47 | 60
  Baseline: Celebrities or social media influencers: Not often or never | 292 | 375
  Baseline: WHO: Often | 170 | 236
  Baseline: WHO: Not often or never | 169 | 199
  Baseline: COVID-19 Hotlines: Often | 144 | 192
  Baseline: COVID-19 Hotlines: Not often or never | 195 | 243
  Baseline: National COVID-19 information website: Often | 163 | 206
  Baseline: National COVID-19 information website: Not often or never | 176 | 229
  Follow-up: Television: Often | 117 | 192
  Follow-up: Television: Not often or never | 222 | 243
  Follow-up: Newspapers: Often | 41 | 49
  Follow-up: Newspapers: Not often or never | 298 | 386
  Follow-up: Health workers: Often | 201 | 289
  Follow-up: Health workers: Not often or never | 138 | 146
  Follow-up: Social media: Often | 76 | 95
  Follow-up: Social media: Not often or never | 263 | 340
  Follow-up: Radio: Often | 70 | 83
  Follow-up: Radio: Not often or never | 269 | 352
  Follow-up: Health department: Often | 193 | 275
  Follow-up: Health department: Not often or never | 146 | 160
  Follow-up: CDC: Often | 167 | 254
  Follow-up: CDC: Not often or never | 172 | 181
  Follow-up: Celebrities or social media influencers: Often | 39 | 56
  Follow-up: Celebrities or social media influencers: Not often or never | 300 | 379
  Follow-up: WHO: Often | 160 | 221
  Follow-up: WHO: Not often or never | 179 | 214
  Follow-up: COVID-19 Hotlines: Often | 130 | 164
  Follow-up: COVID-19 Hotlines: Not often or never | 209 | 271
  Follow-up: National COVID-19 information website: Often | 143 | 181
  Follow-up: National COVID-19 information website: Not often or never | 196 | 254

9. Other Pre Specified Outcome: Trust in Sources of Information
Description: Trust in information sources including television, newspaper, health workers, social media, radio, health department, CDC, hotlines, official websites, and celebrities. (Adapted from the WHO COVID-19 Survey Tool and Guidance).
  "How much do you trust information about COVID-19 from the following sources?"
Time Frame: Baseline and follow-up (4-weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 339 | 435
Participants
  Baseline: Television: Trust | 186 | 269
  Baseline: Television: Little trust or neutral | 153 | 166
  Baseline: Newspapers: Trust | 158 | 160
  Baseline: Newspapers: Little trust or neutral | 181 | 275
  Baseline: Health Workers: Trust | 289 | 388
  Baseline: Health Workers: Little trust or neutral | 50 | 47
  Baseline: Social media: Trust | 104 | 126
  Baseline: Social media: Little trust or neutral | 235 | 309
  Baseline: Radio: Trust | 133 | 164
  Baseline: Radio: Little trust or neutral | 206 | 271
  Baseline: Health Department: Trust | 294 | 386
  Baseline: Health Department: Little trust or neutral | 45 | 49
  Baseline: CDC: Trust | 280 | 375
  Baseline: CDC: Little trust or neutral | 59 | 60
  Baseline: Celebrities and social media influencers: Trust | 57 | 97
  Baseline: Celebrities and social media influencers: Little trust or neutral | 282 | 338
  Baseline: WHO: Trust | 266 | 347
  Baseline: WHO: Little trust or neutral | 73 | 88
  Baseline: COVID-19 Hotlines: Trust | 239 | 314
  Baseline: COVID-19 Hotlines: Little trust or neutral | 100 | 121
  Baseline: National COVID-19 information website: Trust | 243 | 309
  Baseline: National COVID-19 information website: Little trust or neutral | 96 | 126
  Follow-up: Television: Trust | 211 | 272
  Follow-up: Television: Little trust or neutral | 128 | 163
  Follow-up: Newspapers: Trust | 171 | 191
  Follow-up: Newspapers: Little trust or neutral | 168 | 244
  Follow-up: Health workers: Trust | 301 | 371
  Follow-up: Health workers: Little trust or neutral | 38 | 64
  Follow-up: Social media: Trust | 106 | 143
  Follow-up: Social media: Little trust or neutral | 233 | 292
  Follow-up: Radio: Trust | 170 | 179
  Follow-up: Radio: Little trust or neutral | 169 | 256
  Follow-up: Health department: Trust | 290 | 378
  Follow-up: Health department: Little trust or neutral | 49 | 57
  Follow-up: CDC: Trust | 290 | 367
  Follow-up: CDC: Little trust or neutral | 49 | 68
  Follow-up: Celebrities and social media influencers: Trust | 66 | 98
  Follow-up: Celebrities and social media influencers: Little trust or neutral | 273 | 337
  Follow-up: WHO: Trust | 288 | 337
  Follow-up: WHO: Little trust or neutral | 51 | 98
  Follow-up: COVID-19 Hotlines: Trust | 267 | 302
  Follow-up: COVID-19 Hotlines: Little trust or neutral | 72 | 133
  Follow-up: National COVID-19 information website: Trust | 275 | 303
  Follow-up: National COVID-19 information website: Little trust or neutral | 64 | 132

10. Other Pre Specified Outcome: Frequency of Information
Description: Frequency in information. (Adapted from the WHO COVID-19 Survey Tool and Guidance).
Time Frame: Baseline and follow-up (4-weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 339 | 435
Participants
  (Baseline) How often do you seek information about COVID-19?: Often | 88 | 101
  (Baseline) How often do you seek information about COVID-19?: Not often or never | 251 | 334
  (Follow-up) How often do you seek information about COVID-19?: Often | 72 | 102
  (Follow-up) How often do you seek information about COVID-19?: Not often or never | 267 | 333

ADVERSE EVENTS:
Time Frame: 116 weeks
Arm/Group | Intervention | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/517 | 0/534
Serious Adverse Events (participants affected / at risk) | 0/517 | 0/534
Other Adverse Events (participants affected / at risk) | 0/517 | 0/534

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/72/NCT05022472/Prot_003.pdf
  • Statistical Analysis Plan (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/72/NCT05022472/SAP_004.pdf
  • Informed Consent Form (2022-04-04): https://cdn.clinicaltrials.gov/large-docs/72/NCT05022472/ICF_000.pdf